CLINICAL TRIAL: NCT01905774
Title: Renal Function Among Thalassemia Patients Treated by a Oral Chelator Deferasirox
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit, HaEmek Medical Center, Israel
Other Study IDs: 0089-10-EMC
Record Dates: First submitted 2011-09-27; First posted 2013-07-23 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Thalassemia; Iron Overload
Keywords: Renal Function
MeSH Terms: conditions — Thalassemia; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deferasirox: The patients will be treated by the primary physician according to clinical status. The Deferasirox dose range is between 20 to 40 mg/kg/day once daily dose. The treatment is a continuous treatment and not a single course.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox

SUMMARY:
Thalassemia Major patients developed Iron Overload due to blood transfusions and intestinal iron absorption. Renal function caused by Iron overload was studied in a previous study and shows principally tubular disfunction. In this previous study the Iron chelator used was Deferrioxamine. In the last five years an oral Iron chelator was introduced and approved by the FDA, Deferasirox, (Novartis, Switzerland and USA). The purpose of this study is to assess the renal function in Thalassemia Major patients treated with this new oral iron chelator and compare the results with our previous study.

DETAILED DESCRIPTION:
Patients with Thalassemia Major. The laboratory tests that will be studied are: Urine dip stick, Urea, Creatinine, Na, K, Uric Acid, Calcium, Phosphorus in serum and urine, and N acetyl-b-D-glucosaminidase in Urine.Blood gases will be also taken in serum samples.

The overall iron accumulation will also be calculated based in the amount of Packed Cells Units transfused. The total iron burden will also assessed by measurement of Transferrin saturation and Serum Ferritin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Thalassemia Major or Intermedia treated by Iron chelators or by blood transfusions without treatment with iron chelators

Exclusion criteria:

None relevant

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Thalassemia Major or Intermedia treated by Iron chelators or by blood transfusions without treatment with iron chelators
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Renal function in Thalassemia patients treated by Deferasirox | One year study
  Analysis of renal tubular function in patients treated by Deferasirox compared to patients treated by deferrioxamine

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Ha'Emek Medical Center, Afula, Israel

REFERENCES:
- [Background] Smolkin V, Halevy R, Levin C, Mines M, Sakran W, Ilia K, Koren A. Renal function in children with beta-thalassemia major and thalassemia intermedia. Pediatr Nephrol. 2008 Oct;23(10):1847-51. doi: 10.1007/s00467-008-0897-8. Epub 2008 Jun 25. PMID 18581145